CLINICAL TRIAL: NCT04014127
Title: Coronary Microvascular Dysfunction in Chronic Kidney Disease: The Chronic Renal Impairment in Birmingham Coronary Flow Reserve (CRIB FLOW) Study
Brief Title: Coronary Microvascular Dysfunction in Chronic Kidney Disease
Acronym: CRIB-FLOW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Anna Price, Co-Investigator, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK6607
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Kidney Disease, Chronic; Myocardial Dysfunction
Keywords: coronary flow reserve; living kidney donation; peritoneal dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Electrocardiography; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma will be stored for future biomarker analysis including N terminal pro brain natriuretic peptide and troponin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Controls: 25 controls with preserved renal function
  Interventions: Diagnostic Test: Coronary flow reserve assessment; Diagnostic Test: Sphygmocor; Diagnostic Test: Electrocardiogram; Other: Blood test; Other: Urinary albumin/creatinine ratio
- Kidney Donors: 25 living kidney donors who have donated a kidney at least 12 months prior to enrollment in the study.
  Interventions: Diagnostic Test: Coronary flow reserve assessment; Diagnostic Test: Sphygmocor; Diagnostic Test: Electrocardiogram; Other: Blood test; Other: Urinary albumin/creatinine ratio
- Pre-dialysis: 25 patients with pre-dialysis chronic kidney disease stage 5
  Interventions: Diagnostic Test: Coronary flow reserve assessment; Diagnostic Test: Sphygmocor; Diagnostic Test: Electrocardiogram; Other: Blood test; Other: Urinary albumin/creatinine ratio
- Peritoneal dialysis: 25 patients with chronic kidney disease stage 5 undergoing peritoneal dialysis
  Interventions: Diagnostic Test: Coronary flow reserve assessment; Diagnostic Test: Sphygmocor; Diagnostic Test: Electrocardiogram; Other: Blood test; Other: Urinary albumin/creatinine ratio

INTERVENTIONS:
Diagnostic Test: Coronary flow reserve assessment — Coronary flow reserve will be assessed using Doppler transthoracic echocardiograpy and myocardial contrast echocardiography.
Diagnostic Test: Sphygmocor — Pulse wave analysis and pulse wave velocity will be assessed using the Sphygmocor device
Diagnostic Test: Electrocardiogram — An electrocardiogram will be performed prior to administration of adenosine to ensure no resting conduction disease
Other: Blood test — Blood tests will be performed for markers of renal function, bone mineral metabolism and myocardial stretch and injury
Other: Urinary albumin/creatinine ratio — Urine will be analysed for albumin/creatinine ratio

SUMMARY:
This is an observational study assessing coronary microvascular function in healthy controls with normal kidney function, living kidney donors, pre-dialysis patients with chronic kidney disease stage 5 and patients on peritoneal dialysis.

DETAILED DESCRIPTION:
The clinical syndrome of uraemic cardiomyopathy is prevalent in end stage renal disease and is associated with pathological cardiovascular changes including left ventricular hypertrophy, diastolic dysfunction and diffuse interstitial fibrosis. These combine to confer an elevated cardiovascular risk, including an increased risk of sudden cardiac death.

The cause of this increased cardiovascular risk is not clear but it is thought that coronary microvascular dysfunction may play a role. Coronary microvascular dysfunction is prevalent in many myocardial disease states, such as hypertrophic cardiomyopathy and heart failure with preserved ejection fraction, that share pathological similarities with uraemic cardiomyopathy.

Coronary flow reserve, a marker of coronary microvascular function, can be assessed non-invasively using echocardiography techniques. Previous studies have shown a reduction in coronary flow reserve in patients with chronic kidney disease. However, it is not clear if kidney donors - individuals who have a reduced kidney function but do not have progressive kidney disease - also demonstrate microvascular dysfunction. Similarly, although there is some evidence that patients on dialysis have improved coronary flow reserve compared to patients with pre-dialysis chronic kidney disease stage 5, there has been limited investigation into the role of peritoneal dialysis on coronary flow reserve.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control with normal renal function
* Living kidney donor who has donated >12 months prior to enrolment in study
* Chronic kidney disease stage 5 who are pre-dialysis or on peritoneal dialysis
* Able to provide written informed consent

Exclusion Criteria:

* Pregnancy
* Known ischaemic heart disease
* Diabetes mellitus
* Uncontrolled hypertension
* Evidence of 2nd or 3rd degree AV block or sick sinus syndrome in absence of a pacemaker
* History of allergic/adverse reaction to adenosine or Sonovue
* History of long QT syndrome
* Severe hypotension
* Significant valvular heart disease
* Significant chronic obstructive pulmonary disease or asthma with bronchospasm
* Unstable angina not controlled with medication
* Concurrent use of dipyridamole
* Decompensated heart failure
* Poor echo acoustic windows
* Chronic kidney disease stage 5 on haemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending University Hospitals Birmingham.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronary flow reserve | One baseline visit
  Ultrasound-assessed coronary flow reserve. Data will be presented as a ratio (no unit) between maximal mean hyperemia flow velocity and baseline velocity

SECONDARY OUTCOMES:
Myocardial blood flow | One baseline visit
  Ultrasound measurement of myocardial blood flow using myocardial contrast echocardiography. Data will be presented as dB/sec
Left ventricular ejection fraction | One baseline visit
  Echocardiogram assessed left ventricular ejection fraction by Simpson's biplane method. Data will be presented as %.

OTHER OUTCOMES:
Pulse wave analysis | One baseline visit
  Augmentation index measured using the Sphygmocor device. Data will be presented as %.
Pulse wave velocity | One baseline visit
  Pulse wave velocity measured using the Sphygmocor device. Data will be presented as m/s

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Townend, MD FRCP FESC, Principal Investigator — University Hospitals Birmingham
Locations (1):
- Queen Elizabeth Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No